CLINICAL TRIAL: NCT07295899
Title: Evaluation of Impact of Implant Scanning Technique on the Accuracy of Maxillary Complete-arch Digital Scans for Implant-supported Overdentures
Brief Title: Assessing the Influence of Implant Scanning Techniques on the Accuracy of Maxillary Complete-Arch Digital Scans for Implant Overdentures: A Comparative Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Panagiotis Ntovas, PhD Canditate, Department of Operative Dentistry, School of Dentistry, Greece, National and Kapodistrian University of Athens
Other Study IDs: 47/17.07.2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Maxillary Complete-arch Digital Scans for Implant-supported Overdentures
Keywords: Overdenture; Intraoral scanner; Accuracy; Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Scan body (Conventional)
  Interventions: Device: Intraoral scanning
- Scan body (Reverse design)
  Interventions: Device: Intraoral scanning
- Scan body (Apollo design)
  Interventions: Device: Intraoral scanning

INTERVENTIONS:
Device: Intraoral scanning — Different designs of scanbodies will be used

SUMMARY:
Recently different protocols have been developed for the implementation of intraoral scanning in full-arch implant workflows, as horizontal scan body scanning, 1 reverse scanning 2 and scan body systems with an integrated verification jig 3 . The aforementioned approaches are aiming to reduce the inaccuracies related with the implementation of intraoral scanners in full-arch implant cases and to improve the efficiency of the whole digital workflow. However the efficiency of these methods and the parameters that can influence their accuracy, as the design of the scan body have not been investigated.

The purpose of the present in vivo study is to compare the trueness and the precision of the recorded implant's position, between conventional and novel implant acquisition protocols.

DETAILED DESCRIPTION:
The collection of the clinical data for the present research is going to be performed in a private dental clinic.A single patient presenting with an edentulous maxillary arch will be enrolled in the present study.

The patient has to be treated with the placement of four implants and to be planned to be restored with an implant-supported overdenture.In total 3 different scan body systems are going to be evaluated in the present research: conventional scan-bodies (Cares Mono Scan body, Straumann), scan-bodies designed for a horizontal intraoral scanning (Apollo and Reference Scan body, Dynamic abutment), reverse scan bodies (ReveX, Straumann; Scanalog, Dynamic abutment) The scan-bodies will be hand-tightening over the multi-units, which previously will be fixed on 4 implants in patient's maxilla. Each one of the evaluated scan bodies is going to be scanned using an intraoral scanner Trios 5 (3Shape). The verified dentate scan path

recommended by the manufacturer is going to be followed, to scan the reference cast 10 times, for each one of the evaluated scan body systems. The digital scans for each group are going to be performed without removing the scan-bodies in order to eliminate the effect of scan body fit. Finally, an analog impression of splinted impression posts is going to be taken in order to serve as a reference. Based to the analog impression a reference cast is going to be fabricated using a plaster (Type 3, Moldano, Kulzer) and be scanned by a desktop scanner (T710, Medit) using laboratory scan bodies to serve as a reference.The STL files for each evaluated group along with the scans from the industrial scanner will be imported in a metrology software (Geomagic, control X). The digital model derived from each evaluated group is going to be superimposed with the model obtained from the industrial scanner respectively. In order to achieve an accurate superimposition, first "align between measured data" function will be utilized, followed by "best-fit alignment". During the alignment, the area of the scan bodies will be excluded, in order to prevent them from influencing the alignment and the subsequent evaluation. This will be accomplished by using the "use select data only" function. In order to standardize the aforementioned procedure, all superimposed models will be cut simultaneously in the same region.

Afterwards, the overall deviation will be calculated, by using "3D compare" function on Geomagic software, by creating a color map in superimposed digital models to qualitative analyze any 3D deviation. The color map is going to be ranged from -0.5mm to +0.5mm. Mean discrepancy is going to be measured in root mean square RMS, which is a mathematical measure of magnitude of a set of numbers. Trueness will be defined in terms of the mean discrepancy on the positions of the implant abutments, between the digitized by the industrial scanner reference cast and each evaluated group. Precision will be described as the standard deviation of the mean absolute discrepancies computed between the digitized by the industrial scanner reference cast and each evaluated group. A smaller SD indicates that measurements are more precise and consistent, while larger SD will imply greater variability.A power analysis was performed utilizing the G*Power software (G*Power, Heinrich- Heine-Universität Düsseldorf, Germany). The total sample size was calculated based on an effect size of 0.4, an alpha error probability of 0.05, a power of 0.8 and an estimated correlation between measurements of 0.5. The power analysis revealed that a minimum of 10 data sets per evaluated group is required to perform the present study. Statistical analysis will be performed using SPSS statistics software (version 29, IBM software).

Descriptive statistics will be calculated for each evaluated group. The Shapiro-Wilk test will be performed in order to test if the data are normally distributed (P<0.05). For the trueness and the precision, post-hoc analysis (Tukey, Scheffe) will be conducted to assess which evaluated implant acquisition technique will be statistically significantly different.

Fisher's exact test will be used to assess the association between the implant acquisition method and the accuracy of the fit. The level of significance will be set at 0.05. The agreement of fit assessment between the two experienced clinicians will be tested with κ statistics (Cohen's k-score).

ELIGIBILITY:
Inclusion Criteria:

4 implants places in fully edentelous patient that is planned to be treated with implant supported overdenture

-

Exclusion Criteria:

Diseases / Conditions That Can Contraindicate Dental Treatment

1. Uncontrolled Systemic Conditions

   Dental procedures-especially invasive ones-are often postponed if the condition is not medically stable:

   • Uncontrolled Hypertension

   BP typically >180/110 mmHg is considered unsafe for elective dental care.

   Risk: stroke, heart attack during treatment.

   • Uncontrolled Diabetes

   High blood glucose (e.g., >300 mg/dL) increases infection risk and poor healing.

   • Uncontrolled Thyroid Disease

   Hyperthyroidism raises risk of thyroid storm, especially with epinephrine.
2. Recent Major Cardiac Events

   Elective dental treatment is usually deferred for:
   * Heart attack (MI) within past 6 months
   * Stroke within past 6 months
   * Unstable angina
   * Severe arrhythmias
   * Decompensated heart failure

   These conditions can make dental stress or anesthesia dangerous.
3. Infectious Diseases (Active Phase)

   Dental treatment may be delayed to protect the patient or others.
   * Active Herpetic Lesions (Cold Sores) around the mouth
   * Active Tuberculosis (TB)
   * COVID-19 or other acute respiratory infections with fever
4. Hematologic Disorders

   If blood does not clot properly, dental surgery can be risky.

   • Severe Thrombocytopenia

   Platelets too low for safe extraction or surgery.

   • Hemophilia or bleeding disorders

   Require management with a hematologist first.

   • Patients on certain anticoagulants (e.g., warfarin with very high INR)

   May need medical adjustment before invasive care.
5. Pregnancy (Certain Situations)

   Most dental care is safe, but some procedures are postponed:

   Elective treatments during 1st trimester

   Avoid certain medications (e.g., some anesthetics, antibiotics, NSAIDs)

   Severe hypertension or pregnancy complications (eclampsia)
6. Severe Psychiatric Conditions (Unstable)

   When a patient cannot cooperate safely:

   Acute psychosis

   Severe anxiety uncontrolled by medication

   Need medical stabilization vs. dental sedation coordination
7. Substance Intoxication

Dental care is not performed if patient is intoxicated with:

Alcohol

Recreational drugs (especially stimulants like cocaine or meth)

Risk of cardiovascular events or inability to consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental clinical patients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Linear measurements | Through study completion, an average of 1 year, after the execution of all intraoral scans. (Cross-sectional)
  The difference in the linear position between the control and each investigation method would be calculated.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu HK, Wang J, Chen G, Huang X, Deng F, Li Y. Effect of novel prefabricated auxiliary devices attaching to scan bodies on the accuracy of intraoral scanning of complete-arch with multiple implants: An in-vitro study. J Dent. 2023 Nov;138:104702. doi: 10.1016/j.jdent.2023.104702. Epub 2023 Sep 14. PMID 37714453
- [Result] Carneiro Pereira AL, Souza Curinga MR, Melo Segundo HV, da Fonte Porto Carreiro A. Factors that influence the accuracy of intraoral scanning of total edentulous arches rehabilitated with multiple implants: A systematic review. J Prosthet Dent. 2023 Jun;129(6):855-862. doi: 10.1016/j.prosdent.2021.09.001. Epub 2021 Oct 13. PMID 34656307
- [Result] Gomez-Polo M, Donmez MB, Cakmak G, Yilmaz B, Revilla-Leon M. Influence of implant scan body design (height, diameter, geometry, material, and retention system) on intraoral scanning accuracy: A systematic review. J Prosthodont. 2023 Dec;32(S2):165-180. doi: 10.1111/jopr.13774. Epub 2023 Oct 18. PMID 37771200
- [Result] Revilla-Leon M, Smith Z, Methani MM, Zandinejad A, Ozcan M. Influence of scan body design on accuracy of the implant position as transferred to a virtual definitive implant cast. J Prosthet Dent. 2021 Jun;125(6):918-923. doi: 10.1016/j.prosdent.2020.03.019. Epub 2020 May 31. PMID 32493568
- [Result] Papaspyridakos P, Bedrossian A, Kudara Y, Ntovas P, Bokhary A, Chochlidakis K. Reverse scan body: A complete digital workflow for prosthesis prototype fabrication. J Prosthodont. 2023 Jun;32(5):452-457. doi: 10.1111/jopr.13664. Epub 2023 Mar 3. PMID 36779654
- [Result] Giglio GD, Giglio AB, Tarnow DP. A Paradigm Shift Using Scan Bodies to Record the Position of a Complete Arch of Implants in a Digital Workflow. Int J Periodontics Restorative Dent. 2024;44(1):115-126. doi: 10.11607/prd.6733. PMID 37552170